CLINICAL TRIAL: NCT04695353
Title: Study of Feasibility and Efficacy of Telecommunication Platforms as an Adjunctive Clinical Tool for a Parkinson's Disease Clinic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario de Burgos (Other)
Responsible Party: Principal Investigator, Esther Cubo, MD, PhD, Principal Investigator, Hospital Universitario de Burgos
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: CEIC-2299
Record Dates: First submitted 2020-12-30; First posted 2021-01-05 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Parkinson Disease
Keywords: telemedicine; Cost-effectiveness
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: International, longitudinal, case-control study comparing in-office visits to virtual visits via Telecommunication Platforms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): These patients will receive telemedicine by using Telecommunication Platform videoconferences/messages.
  Interventions: Procedure: Telemedicine: Virtual visits (videoconferences, texts)
- Control group (No Intervention): The patients will receive in-office clinical care

INTERVENTIONS:
Procedure: Telemedicine: Virtual visits (videoconferences, texts) — Patients will receive clinical care by using telemedicine (virtual visits)
  Arms: Study group

SUMMARY:
Telecommunication Platforms are new technology founded to build better short messages service alternative. Their use have increasingly drawn a wider range of interest as a text communication and video chat system between health care professionals and patients and health care professionals themselves. However, high-quality and adequately evaluated research, especially in the field of neurodegenerative diseases such as Parkinson´s disease, is needed to establish whether patients with these specific neurological problems can be effectively managed with these technological tools in low, middle, and high-income countries

DETAILED DESCRIPTION:
Telecommunication Platforms are new technology founded to build a better short message service alternative. Their use have increasingly drawn a wider range of interest as a text communication and video chat system between health care professionals and patients and health care professionals themselves. However, high-quality and adequately evaluated research, especially in the field of neurodegenerative diseases such as Parkinson´s disease, is needed to establish whether patients with these specific neurological problems can be effectively managed with these technological tools. In this study, patients with Parkinson´s disease from high, middle, and low-income countries covering urban and rural populations, with at least one neurologist with Movement Disorders practice (Spain, Uruguay, Saudi Arabia, Nigeria, Tanzania, South Korea, United States, Egypt), will be included. Feasibility, clinical management, providers and patient´s satisfaction will be compared between in-office vs. telemedicine (virtual) visits. This study will show the effectiveness of telemedicine, when the access to specialized neurological care is limited, especially now with the Covid-19 pandemic.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with idiopathic Parkinson´s disease, able to use a smart phone and running videoconferences, with easy access to wifi.

Exclusion Criteria:

Patients with severe ambulatory problems that will interfere with in-office visits, without access to Internet, with limited technical knowledge unable to use Telecommunication Platforms, or patients diagnosed with other types of Parkinsonism.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-02-28 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of Virtual Visits for Parkinson Disease | 1 year
  number of scheduled in-office and virtual visits that are completed, overall as well as by center, gender, and age-group.
Clinical management Complexity | 1 year
  Comparison of the clinical issues frequency (% of any of the following) performed during either virtual or in-office visits: the sum of pharmacological and non-pharmacological treatment recommendations, urgent clinical problem evaluation, discussion of test results, education, and second-opinion requests
Patients and providers satisfaction and difficulties | 1 year
  description and comparison of the main difficulties and overall satisfaction between virtual vs. in-office visits

SECONDARY OUTCOMES:
Cost-effectiveness | 1 year
  Comparison of costs (from a patient's perspective) at the end of the study vs. baseline (previous 6 months) in terms of medical (drugs, doctors and other health professionals, hospitalizations, non-pharmacological interventions, work-up tests), and non-medical (internet and cellular phone fee, travel costs related to health care, medical equipments such as canes, etc, caregiver and nursing home fees) costs between virtual and in-office visits

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario de Burgos, Burgos, Spain

IPD SHARING:
Plan to Share IPD: No